CLINICAL TRIAL: NCT04881916
Title: Elucidating Novel Immune and Genomic Markers for ALK (ENIGMA+)
Brief Title: Immune and Genomic Markers in ALK+ NSCLC
Status: Active, not recruiting | Type: Observational
Sponsor: Massachusetts General Hospital (Other)
Collaborators: LUNGevity Foundation (Other); Addario Lung Cancer Medical Institute (Other)
Responsible Party: Principal Investigator, Jessica Jiyeong Lin, M.D., Principal Investigator, Massachusetts General Hospital
Other Study IDs: 20-237
Record Dates: First submitted 2021-05-06; First posted 2021-05-11 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-08

CONDITIONS: Anaplastic Lymphoma Kinase Gene Translocation; Non-Small Cell Lung Cancer
Keywords: Anaplastic Lymphoma Kinase Gene Translocation; Non-Small Cell Lung Cancer; ALK
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Biospecimen Retention: Samples With DNA — Tissue and saliva specimens
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Sample Collection: Participation In:
  * Initial data completion: Telephone collection of information on disease, treatment and testing
  * Medical record collection: Collection of medical records regarding cancer, testing, and treatment history
  * Archival tissue collection: Collection of tumor from prior standard of care procedure
  * Saliva collection: Saliva collection with at home kit
  * Follow up data completion: Telephone collection of medical condition every 3-6 months up to 2 years.

SUMMARY:
The purpose of this research study is to obtain and study clinical history, and tissue and saliva specimens if available from participants with Anaplastic Lymphoma Kinase-ALK+ Non-Small Lung Cancer(NSCLC)

DETAILED DESCRIPTION:
The purpose of this study is to establish a registry of clinical data and tumor specimens of patients with advanced ALK+ non-small lung cancer (NSCLC) (defined as NSCLC harboring an ALK gene rearrangement). This will allow in-depth, comprehensive genomic and immunophenotypic analyses of ALK+ tumors. Together with the clinical data, these biologic specimens will enable the conduct of basic and translational research to identify genomic and immunologic markers associated with clinical outcomes for ALK+ patients.

ELIGIBILITY:
Inclusion Criteria:

Cohort 1 - Alive Individuals

* Men or women 18 years of age or the age of majority for their residential state of the United States, or older, at the time of consent.
* Histologically or cytologically confirmed advanced stage IIIB-IIIC not amenable to curative approach multi-modality (e.g., chemoradiation and/or surgery) treatment, or stage IV non-small cell lung cancer (NSCLC)
* Demonstration of having advanced ALK+ NSCLC, as assessed by fluorescence in situ hybridization (FISH), immunohistochemistry (IHC), next-generation sequencing (NGS) or circulating tumor DNA analysis (ctDNA). For ALK FISH, fusions must have been detected in at least 15% of tumor cells.
* Willingness to provide clinical and medical information to the study team as required.
* Willingness to provide archival tumor tissue, if available. Patients may enroll even if no tumor tissue is available.
* Ability to read, write and communicate in English.
* Ability to sign a web-based informed consent form.

Cohort 2 - Deceased Individuals

* Deceased individuals diagnosed with advanced ALK+ lung cancer at age 18 years or older may be studied on a case by case basis. Inclusion will require availability of adequate archived tissue and release of tissue and records by next of kin, if available.

Exclusion Criteria:

* Participants who are unwilling to provide informed consent.
* Participants who are younger than 18 years of age.
* Participants who are unable to comply with the study procedures.
* Known existence of an uncontrolled intercurrent illness including, but not limited to, psychiatric illness or social situations that would impair compliance with study requirements.
* Participants who have previously enrolled to the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with advanced ALK-positive (ALK+) non-small cell lung cancer (NSCLC)
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-12-01 (Actual); Primary Completion 2027-07-01 (Estimated); Study Completion 2027-07-01 (Estimated)

PRIMARY OUTCOMES:
Registry Establishment | Up to 2 years
  Establish a registry of clinical data and tumor specimens from goal of 100 patients with advanced ALK+ NSCLC (defined as NSCLC harboring an ALK gene rearrangement), for characterization of the immunophenotype and genomic landscape of ALK+ NSCLC.

SECONDARY OUTCOMES:
Duration Of Therapy | Up to 2 years
  To determine the clinical outcomes (durations of therapy) on ALK Tyrosine kinase inhibitor-TKI(s) and/or immune checkpoint inhibitor-ICI(s) of ALK+ NSCLC patients. Duration of therapy will be estimated using the Kaplan-Meier method, and 95% confidence intervals (CIs) will be calculated using the log-log transformation.
Overall survival (OS) | Up to 2 years
  To determine the overall survival (OS) of ALK+ NSCLC patients treated with sequential ALK TKIs and/or ICIs. OS for patient will be estimated using the Kaplan-Meier method, and 95% confidence intervals (CIs) will be calculated using the log-log transformation Overall survival (OS) will be calculated as the time from the first dose of the drug of interest to death due to any cause.
ALK resistance mutations | Up to 2 years
  Study the development of ALK resistance mutations in the TKI-resistant tumor specimen(s) as patients receive sequential ALK-targeted therapies
Genomic alterations | Up to 2 years
  To determine the presence of genomic alterations such as single nucleotide variants, insertions or deletions, or copy number alterations in other cancer-related genes in the post-TKI tumor specimen(s).
Tumor immunophenotype | Up to 2 years
  Correlate the tumor immunophenotype such as PD-L1 expression level or tumor mutational burden (TMB) with clinical outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Jessica J Lin, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital Cancer Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to: [contact information for Sponsor Investigator or designee]. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact the Partners Innovations team at http://www.partners.org/innovation

REFERENCES:
- [Derived] Liang J, Waliany S, Do A, Peterson JL, Roberts P, Kennedy EA, Venanzi ES, Gainor JF, Lin JJ. ENIGMA+: a national, decentralized, remote consent study for clinical data and biospecimen collection in patients with ALK-positive advanced NSCLC. Oncologist. 2025 Sep 1;30(9):oyaf217. doi: 10.1093/oncolo/oyaf217. PMID 40674592